CLINICAL TRIAL: NCT00116129
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of MK-0677 25 mg in the Treatment of Primary Fibromyalgia
Brief Title: Efficacy and Safety of an Oral Growth Hormone Drug in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bennett, Robert, M.D. (Individual)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Robert Bennett MD, Professor of Medicine OHSU, Bennett, Robert, M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MK-0677/FM; IND 71,596
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Treatment; Growth hormone; IGF-1; MK-0677; Oral growth hormone secretagogue
MeSH Terms: conditions — Fibromyalgia | interventions — ibutamoren mesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Ibutamoren Mesylate (MK-0677)

INTERVENTIONS:
Drug: Ibutamoren Mesylate (MK-0677) — Ibutamoren Mesylate 25 mg/day

SUMMARY:
This is a 24-week, randomized, double-blind, placebo-controlled, trial to evaluate the safety, tolerability and efficacy of an orally administered growth hormone stimulating drug, (code named MK-0677) in the treatment of female subjects with primary fibromyalgia. The basis for this study is the observation that many fibromyalgia patients are growth hormone deficient; an earlier study of injectable growth hormone had shown benefit in this population of fibromyalgia patients.

DETAILED DESCRIPTION:
This study examines whether MK-0677 treatment will improve symptoms of fibromyalgia (FM).

The rationale for this study is the observation that many fibromyalgia patients are growth hormone deficient in terms of low levels of IGF-1, and that improving IGF-1 levels with growth hormone injections has been shown to improve fibromyalgia symptoms.

MK-0677 is an orally administered growth hormone secretagogue manufactured by Merck & Co., Inc. that acts on the growth hormone secretagogue receptor in the anterior pituitary to stimulate the release of growth hormone. This pathway represents an additional regulation of growth hormone release from pituitary somatotrophs to that mediated by growth hormone releasing hormone (stimulating) and somatostatin (inhibitory). Both stimulatory pathways lead to a pulsatile release of growth hormone, with approximately 4 hour intervals between peak levels. This growth hormone secretion leads to a rapid and robust up regulation of IGF-1 levels by about 50 to 100% that can be maintained with chronic therapy at a dose of 25 mg/day.

The primary aims of this study are:

1. To evaluate the efficacy of MK-0677 25 mg in primary fibromyalgia subjects over a 24-week treatment period, as assessed by the FIQ.
2. To evaluate the safety and tolerability of MK-0677 25 mg in subjects with fibromyalgia.

The secondary aims of this study are to determine whether:

1. MK-0677 25 mg is superior to placebo in reducing muscle tenderness, as assessed by the Fibromyalgia Myalgic Score (FMyS).
2. MK-0677 25 mg is superior to placebo in improving the subjects' global perception of change in fibromyalgia symptoms, as assessed by the Subjects' Global Impression of Change Questionnaire (PGIC).
3. MK-0677 25 mg is superior to placebo in improving the subjects' quality of life, as assessed by the Quality of Life Questionnaire (QOL).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will all be female primary fibromyalgia subjects who are 30 to 65 years of age, inclusive, and have a low age adjusted serum IGF-1 level.
* All subjects will fulfill a diagnosis of fibromyalgia according to the classification criteria of the American College of Rheumatology (ACR).
* All subjects will have an initial Fibromyalgia Impact Questionnaire (FIQ) score ≥ 40.
* If subject is of childbearing potential and sexually active, she agrees to use effective barrier or appropriate oral contraception during the study. Subjects who are taking oral contraceptives must have done so for at least 2 months prior to entering the study.
* Subject is not pregnant and is not nursing.
* Patient has a normal screening breast exam. If screening breast exam is abnormal, but not suggestive of breast cancer, the patient must have had a normal mammogram within the last 6 months.
* Subject has a normal screening stool hemoccult. If the screening stool hemoccult is abnormal, but likely due to hemorrhoids, the subject must have had a normal sigmoidoscopy within the last 2 years.
* Subject is willing to discontinue using grapefruit juice for duration of study.
* Subject is willing to be followed by telephone contact for 3 months after she has discontinued study and completed and returned the Fibromyalgia Impact Questionnaire, Patient Global Change score, Quality of Life score, Brief Pain Inventory and Beck Depression Questionnaire.

Exclusion Criteria:

* Subject has an-ongoing, unresolved disability litigation.
* Subject has diabetes or a significantly elevated random glucose at the Screening visit.
* Subject has a current or past history of cardiovascular, pulmonary, neurological, endocrine or renal disease that would preclude involvement in an exercise program (specifically hypertension, a myocardial infarction within the last 6 months, chronic obstructive pulmonary disease [COPD], asthma, untreated hypothyroidism, severe depression with suicide risk, previous pituitary disease or surgery).
* Subject has a history of angina or congestive heart failure with symptoms that occur at rest.
* Subject has a history or current evidence of a psychotic disorder (e.g. schizophrenia), bipolar disorder or major depression, or substance abuse by DSM-IV criteria; severe depression, as evidenced by a Beck Depression score of ≥ 30.
* Subject has history of neurological disorder other than fibromyalgia (e.g. epilepsy, stroke, neuropathy, neuropathic pain).
* Subject has ongoing symptoms of carpal tunnel syndrome.
* Subject has any other significant pain state, i.e. subject must have primary fibromyalgia.
* Subject has a history of hepatitis or liver disease that has been active within the past 12 weeks.
* Subject has cancer or a history of cancer within the past 2 years, or a history of cancer of more than 2 years ago and deemed to not be cured, or subject has ANY history of breast cancer. (NOTE: Subjects with a history of basal cell or squamous cell carcinoma of the skin treated more than 1 year ago and with no evidence of recurrence may participate.)
* Subject has abnormal thyroid stimulating-hormone, or T4 concentrations.
* Subject has a planned elective surgery during the study period.
* Subject has a history of hypersensitivity or idiosyncratic reaction to more than 2 drug classes (by chemical classification).
* Subject has abnormal Screening visit laboratory values.
* Subject is using any of the following medications : heparin, ticlopidine, ginko (in subjects taking warfarin), oral steroids (>/= 7 days per month), chronic use of strong CYP3A4 inhibitors (HIV protease inhibitors, macrolide antibiotics and nefazodone), chronic use of CYP3A4 inducers (carbamazepine, phenytoin, rifampin, and St. John's Wort).

  p. Subject has received an investigational drug or device within 30 days of study entry.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
MK-0677 25 mg is superior to placebo in reducing symptoms of fibromyalgia, as assessed by the Fibromyalgia Impact Questionnaire (FIQ) over a 24-week treatment period | Six months
MK-0677 25 mg is generally safe and well tolerated in subjects with fibromyalgia | Six months

SECONDARY OUTCOMES:
MK-0677 25 mg is superior to placebo in improving the subjects' global perception of change in fibromyalgia symptoms, as assessed by the Subjects' Global Impression of Change Questionnaire (PGIC) | Six months
MK-0677 25 mg is superior to placebo in improving the subjects' quality of life, as assessed by the Quality of Life Questionnaire (QOL) | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bennett, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Bennett RM, Cook DM, Clark SR, Burckhardt CS, Campbell SM. Hypothalamic-pituitary-insulin-like growth factor-I axis dysfunction in patients with fibromyalgia. J Rheumatol. 1997 Jul;24(7):1384-9. PMID 9228141
- [Background] Bennett RM, Clark SC, Walczyk J. A randomized, double-blind, placebo-controlled study of growth hormone in the treatment of fibromyalgia. Am J Med. 1998 Mar;104(3):227-31. doi: 10.1016/s0002-9343(97)00351-3. PMID 9552084